CLINICAL TRIAL: NCT01761292
Title: A Two-Part Study to Assess the Safety and Tolerability, Pharmacokinetics, and Effects on Histology and Different Clinical Parameters of Givinostat in Ambulant Children With Duchenne Muscular Dystrophy
Brief Title: A Study to Assess Safety/Tolerability, pk, Effects on Histology, Clinical Parameters of Givinostat in Children With DMD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/11/2357/43; 2012-002566-12 (EudraCT Number)
Record Dates: First submitted 2012-12-20; First posted 2013-01-04 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2020-06

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: rare disease
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Rare Diseases | interventions — givinostat; givinostat hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Givinostat (Experimental): Givinostat will be administered as 2 oral doses daily while the child is in fed state.
  Interventions: Drug: Givinostat

INTERVENTIONS:
Drug: Givinostat — Givinostat, oral suspension 10 mg/mL or oral capsules 50 mg, administered orally under fed conditions at the dose of 25 mg BID, 37.5 mg BID, and 50 mg BID during Part 1 for two weeks, and 25 mg BID and 37.5 mg BID during Part 2 for 12 months. Givinostat, oral suspension 10 mg/mL, administered orally under fed conditions at the dose of 25 mg BID or 37.5 mg BID during Extension 1, and modified as per patient's weight during Extensions 2 and 3 (up to 52 months).
  Other Names: ITF2357

SUMMARY:
The primary objective of Parts 1 and 2 of the study were to establish the histologic effects of givinostat administered chronically at the selected daily dose.

The secondary objectives of Parts 1 and 2 of the study were as follows:

* To establish the effects of givinostat administered chronically at the selected daily dose on functional parameters, such as the 6-Minute Walk Test (6MWT), North Star Ambulatory Assessment (NSAA), and performance of upper limb (PUL)
* To establish the safety and tolerability of givinostat administered chronically at the selected daily dose in children with Duchenne muscular dystrophy (DMD)
* To explore the effects of givinostat administered chronically at the selected daily dose on parameters such as magnetic resonance imaging (MRI) and biomarkers
* To explore the acceptability/palatability of the oral suspension
* To explore whether the effects of givinostat on disease progression may be related to the type of DMD mutation.

The primary objective of the Extension of the study was to evaluate the safety and tolerability of long-term administration of givinostat administered chronically at the selected daily dose in children with DMD.

The secondary objectives of the Extensions were:

* To establish the effects of givinostat administered chronically at the selected daily dose on muscular functional parameters, such as the 6MWT, NSAA, and PUL (Extensions 1, 2, and 3)
* To explore the effects of givinostat administered chronically at the selected daily dose on parameters such as MRI (Extension 1)
* To collect information related to 2 biomarkers, latent Transforming growth factor β (TGFβ) binding protein 4 (LTBP4) and osteopontin genotype (at the beginning of Extension 2 only)
* To collect information related to time to wheelchair and how much time the children spend in wheelchair (Extension 3 - only for the children who were not able to complete the 6MWT)

DETAILED DESCRIPTION:
This is a 2-part, phase II study to assess the effects of Givinostat on muscle histologic parameters and on clinical parameters in ambulant children with DMD.

The safety, tolerability, and pharmacokinetics of Givinostat will also be assessed.

Approximately 20 children were to be enrolled in the study as follows: the first 4 children were to be treated at a low dose level of givinostat (25 mg twice daily [BID] in children who weighed 20 kg to 49 kg and 37.5 mg BID in children who weighed ≥ 50 kg).

If none of the stopping criteria were met after 2 weeks of treatment at the low dose, the review team was to determine the escalated dose level (ie, intermediate dose level) to be used for the treatment of an additional 8 children who were to be treated at the intermediate dose. The 4 children previously treated at the low dose level were also switched to the intermediate dose level.

If none of the stopping criteria were met after 2 weeks of treatment at the intermediate dose, the review team was to determine the subsequent escalated dose level to be used for the treatment of an additional 8 children who were to be treated at the high dose. All children treated at the intermediate dose level were to be switched to the high dose level.

Once all 20 children enrolled during Part 1 of the study had been treated for at least 2 weeks, the review team was to determine the recommended dose (RD) to be used in Part 2 based on the safety and tolerability profile observed and on the pharmacokinetic (PK) analyses. All the children enrolled were switched to the RD level (37.5 mg BID), which was administered for the subsequent 12 months of the study (Part 2).

At the end of Part 2 of the study, parents were asked to consent and patients to assent to continuing their participation in the Extension to receive the study treatment at least until the final analysis was performed (Part 3-Extensions; after 52 months of treatment). The patients received givinostat at the same ongoing dose, during the last visit planned at 12 months, and were treated for additional 40 months (Extensions 1, 2, and 3 up to month 52).

ELIGIBILITY:
Inclusion Criteria:

1. Male children aged 7 to <11 years with an immunohistochemical and molecular diagnosis of DMD.
2. A parent/guardian and child can comply with all study evaluations/procedures and return for all study activities.
3. Able to complete the 2 screening 6MWTs with a minimal distance of at least 250 m each. In addition, the results of these tests must be within ±30 m of each other.
4. On a stable dose of systemic corticosteroids for at least 6 months.
5. At least 6 months worth of data on the 6MWT (this will be the "historical" 6MWT). From the moment of the historical 6MWT assessment(s), the child must not have received any compound that could potentially affect the 6MWT, with the exception of the stable steroid treatment.
6. Parent/guardian has signed the informed consent form and child has assented to be in the study (if applicable).

Exclusion Criteria:

1. Initiation of systemic corticosteroid therapy within 6 months prior to the start of study drug or change in systemic corticosteroid therapy (e.g., initiation, change in type of drug, dose modification not related to body weight change, schedule modification, interruption, discontinuation, or re initiation) within 6 months prior to the start of study drug.
2. Use of any pharmacologic treatment, other than corticosteroids, that might have an effect on muscle strength since the time of the historical 6MWT and in any case within 3 months prior to the start of study treatment (e.g., growth hormone). Vitamin D, calcium, and integrators will be allowed.
3. Surgery that might have an effect on muscle strength or function within 3 months before study entry or planned surgery at any time during the study.
4. Exposure to another investigational drug since the time of the historical 6MWT and in any case within 3 months prior to the start of study treatment.
5. History of participation in gene therapy, cell-based therapy or oligonucleotide therapy.
6. Presence of other clinically significant disease that in the opinion of the investigator places the child in unacceptable risk for an adverse outcome or that could affect study results.
7. Symptomatic cardiomyopathy or heart failure. If child has a left ventricular ejection fraction <45% at screening, the investigator should discuss inclusion of child in the study with the medical monitor.
8. Inadequate hematological function
9. Absolute neutrophil count: <1.5 x 109/L
10. Platelets: <100 x 109/L
11. Current or history of liver disease or impairment, including but not limited to an elevated total bilirubin.
12. Inadequate renal function, as defined by serum creatinine >2 x the upper limit of normal.
13. Positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus at screening
14. A baseline QTc >450 msec, (as the mean of 3 consecutive readings 5 minutes apart) or history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome).
15. Psychiatric illness/social situations rendering the potential child unable to understand and comply with the study protocol.

Ages: 7 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Bertini, MD, Principal Investigator — Bambino Gesù Children's Hospital, IRCCS, Rome, Italy.
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Policlinico Agostino Gemelli, Roma
  - Ospedale Pediatrico Bambino Gesù, Rome

REFERENCES:
- [Result] Bettica P, Petrini S, D'Oria V, D'Amico A, Catteruccia M, Pane M, Sivo S, Magri F, Brajkovic S, Messina S, Vita GL, Gatti B, Moggio M, Puri PL, Rocchetti M, De Nicolao G, Vita G, Comi GP, Bertini E, Mercuri E. Histological effects of givinostat in boys with Duchenne muscular dystrophy. Neuromuscul Disord. 2016 Oct;26(10):643-649. doi: 10.1016/j.nmd.2016.07.002. Epub 2016 Jul 11. PMID 27566866

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a single arm study and not a parallel group study. Patient enrollment occurred sequentially, until 20 patients were treated (part 1). For the entire design please refer to "detailed study description". Only demographics are reported by 3 Givinostat dose levels, while AEs and outcomes results are reported for the whole Givinostat population.
Groups:
- Givinostat: Givinostat will be administered as 2 oral doses daily while the child is in fed state.
  Givinostat: Givinostat, oral suspension 10 mg/mL or oral capsules 50 mg, administered orally under fed conditions at the dose of 25 mg BID, 37.5 mg BID, and 50 mg BID during Part 1 and 25 mg BID and 37.5 mg BID during Part 2. Givinostat, oral suspension 10 mg/mL, administered orally under fed conditions at the dose of 25 mg BID or 37.5 mg BID during Extension 1, and modified as per patient's weight during Extensions 2 and 3.
Period: Part 1
Arm/Group | Givinostat
Started | 20
Patients Receiving Drug in Part 1 | 19 (One patient was enrolled in Part 1 and started treatment in Part 2.)
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — not receiving treatment in Part 1 | 1
Period: Part 2
Arm/Group | Givinostat
Started | 19 (1 pt was enrolled in Part 1 but started the treatment in Part 2. So 19 pts started Part 2.)
Completed | 19
Not Completed | 0
Period: Extension 1
Arm/Group | Givinostat
Started | 19
Completed | 18
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Extension 2
Arm/Group | Givinostat
Started | 18
Completed | 18
Not Completed | 0
Period: Extension 3
Arm/Group | Givinostat
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The ITT population included all children who were enrolled in the Part 1 portion or entered the Part 2 portion of the study. Patients were analyzed according to the dose level to which they were allocated. Twenty patients were included in the ITT population.
Groups:
- ITF2357 25 mg BID: Givinostat, oral suspension 10 mg/mL, administered orally under fed conditions at the dose of 25 mg BID, during Part 1 and 25 mg BID during Part 2 and during Extension 1.
  The dosage was modified as per patient's weight during Extensions 2 and 3.
- ITF2357 50 mg BID: Givinostat oral capsules 50 mg, administered orally under fed conditions at the dose of 50 mg BID during Part 1.
  The dosage was modified as per patient's weight during Extensions 2 and 3.
- ITF2357 37.5 mg BID: Givinostat, oral suspension 10 mg/mL, administered orally under fed conditions at the dose of 37.5 mg BID during Part 1 and 37.5 mg BID during Part 2 and during Extension 1.
  The dosage was modified as per patient's weight during Extensions 2 and 3.
- Total: Total of all reporting groups
Arm/Group | ITF2357 25 mg BID | ITF2357 50 mg BID | ITF2357 37.5 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 8 | 8 | 20
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (0.96) | 8.8 (1.16) | 7.9 (1.13) | 8.2 (1.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 8 | 8 | 20
Region of Enrollment [Number; unit: participants]
  Italy | 4 | 8 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Part 2 in the Value of Muscle Fiber Area (MFA) % Comparing the Histology Biopsies Before and After 12 Months of Treatment With Givinostat.
Description: The primary endpoint was the change in histology comparing the brachial biceps biopsies before and after ≥12 months of treatment with Givinostat.
  Muscle biopsies: A first brachial biceps biopsy (baseline) was taken prior to the first dose of study drug. A second brachial biceps biopsy was taken at Visit 10 (12 months) from the opposite arm.
  The muscle biopsy samples from the biceps muscle were collected by open biopsy. The minimum amount of muscle tissue required was a piece of muscle of at least 0.5 × 0.5 × 0.5 cm.
Time Frame: After12 months of treatment
Population: Evaluable population:all patients who received givinostat of at least 80% dose in Part 2, had at least 1 baseline and 1 post baseline biopsy and no major protocol violations. 19 Subjects completed Part 2, 1 subject was excluded by this analysis due to biopsy not readable. Results data are reported only for the "overall" Givinostat population.
Measure: Median (Full Range); unit: percentage change
Groups:
- Overall: Givinostat was administered as 2 oral doses daily while the child is in fed state.
  Givinostat, oral suspension 10 mg/mL or oral capsules 50 mg, was administered at the dose of 25 mg BID, 37.5 mg BID, and 50 mg BID during Part 1, and 25 mg BID and 37.5 mg BID during Part 2.
Arm/Group | Overall
Number analyzed (Participants) | 18
percentage change | 12.76 [6.17 to 21.23]
Statistical Analysis 1: Comparison: Overall; Test type: Other; p < 0.0001, t-test, 2 sided — The paired t-test or non-parametric signed rank test for 2 means (paired observations) (as is appropriate) was applied for testing the statistical significance of the Change From Baseline to End of Study. MFA% P < 0.05 was set as significant; mean = 13.906, 95% CI 2-sided [11.5657 to 16.2466]

2. Secondary Outcome: Change From Baseline to End of Study in Cross Sectional Area (CSA)
Description: This histological parameter was evaluated on the brachial biceps biopsies taken prior to the first dose of study drug and after 12 months of treatment with givinostat.
Time Frame: At 12 months
Population: The ITT population included all children who were enrolled in the Part 1 or entered the Part 2 of the study. For histology parameters patients were analyzed "overall" for Givinostat population. 19 completed part 2 but only 18 subejcts had 2 biopsies readable
Measure: Mean (Standard Deviation); unit: μm2
Arm/Group | Overall
Number analyzed (Participants) | 18
μm2 | 865.269 (555.3543)
Statistical Analysis 1: Comparison: Overall; Test type: Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Change From Baseline to End of Study in Fibrosis, Necrosis, Fatty Replacement
Description: These histological parameters were evaluated on the brachial biceps biopsies taken prior to the first dose of study drug and after 12 months of treatment with givinostat.
Time Frame: After 12 months
Population: The ITT population included all children who were enrolled in the Part 1 or entered the Part 2 of the study. For histology parameters patients were analyzed "overall" for Givinostat population. 19 Subjects completed Part 2 but only 18 had 2 biopsies readable.
Measure: Mean (Standard Deviation); unit: percentage of total area
Groups:
- Baseline: Givinostat was administered as 2 oral doses daily while the child is in fed state.
  Givinostat, oral suspension 10 mg/mL or oral capsules 50 mg, was administered at the dose of 25 mg BID, 37.5 mg BID, and 50 mg BID during Part 1, and 25 mg BID and 37.5 mg BID during Part 2.
Arm/Group | Baseline
Number analyzed (Participants) | 18
percentage of total area
  Total fibrosis | -12.640 (4.6493)
  Perimysial fibrosis | -7.585 (6.4779)
  Endomysial fibrosis | -5.056 (6.2531)
  Fatty replacement | -0.302 (0.2756)
  Necrosis | -0.964 (0.6260)

4. Secondary Outcome: Change From Baseline to End of Study in Number of Hypercontracted Fibers
Description: This histological parameter was evaluated on the brachial biceps biopsies taken prior to the first dose of study drug and after 12 months of treatment with givinostat. The number of fibers is calculated per microscopic field (20x).
Time Frame: At 12 months
Population: The ITT population included all children who were enrolled in the Part 1 or entered the Part 2 of the study. For histology parameters patients were analyzed "overall" for Givinostat population.19 Subjects completed Part 2 but only 18 had 2 biopsies readable.
Measure: Mean (Standard Deviation); unit: number of fibers
Arm/Group | Overall
Number analyzed (Participants) | 18
number of fibers | -1.204 (0.6621)

5. Secondary Outcome: Change From Baseline in Muscular Function After 12 Months of Treatment With Givinostat at the Selected Daily Dose Based on the 6-Minute Walk Test
Description: This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
  The 6-Minute Walk Test is a useful measure of functional capacity targeted at people with at least moderately severe impairment.
  The longer the walked distance the better the outcome.
Time Frame: At 12 months
Population: The ITT population included all children who were enrolled in the Part 1 portion or entered the Part 2 portion of the study. Results data are reported only for the "overall" Givinostat population, due to a small sample. 19 subjects completed Part 2 of the study 19 but only 18 performed the 6-Minute Walk Test
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Overall
Number analyzed (Participants) | 18
meters | -24.6 (36.11)

6. Secondary Outcome: Change From Baseline in Muscular Function After 12 Months of Treatment With Givinostat at the Selected Daily Dose Based on the North Star Ambulatory Assessment (NSAA)
Description: The NSAA, which is composed by 17 items, was graded, for each item, using the standard scorecard with each assessment rated as 0 - unable to achieve independently, 1 - modified method but achieves goal independent of physical assistance from another, or 2 - normal with no obvious modification of activity.
  The subscales scores are summed up to compute a total score, ranging from 0 to 34. The higher the total score, the better the outcome.
  The mean Change From Baseline to EoS in NSAA total score is reported hereunder.
Time Frame: At 12 months
Population: The ITT population included all children who were enrolled in the Part 1 portion or entered the Part 2 portion of the study. Patients were analyzed "overall" due to a small sample size. Although different Givinostat dose levels were administered, results data are reported only for the "overall" Givinostat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall
Number analyzed (Participants) | 19
score on a scale | -2.8 (3.15)

7. Secondary Outcome: Change From Baseline in Muscular Function After 12 Months of Treatment With Givinostat at the Selected Daily Dose Based on the Performance of Upper Limb (PUL)
Description: The PUL (version 1.2) was used to assess the change in motor performance of the upper limb over time in patients with Becker and Duchenne muscular dystrophy, from when they are still ambulant, until they loose all arm function when non-ambulant.
  The revised version of the PUL included 22 items. These include one entry item to define the starting functional level, and 21 items subdivided into:
  * shoulder level (Question B to E; minimum score 0 and maximum score 16)
  * elbow level (Question F to N; minimum score 0 and maximum score 34)
  * distal level dimension (Question O to V; minimum score 0 and maximum score 24) The total score is calculated by the sum of all the scores of the three subscales (total score range: 0-74) (scores from Question A "entry item" did not contribute). For all items, the higher the score, the better the outcome.
Time Frame: At 12 months
Population: The ITT population included all children who were enrolled in the Part 1 portion or entered the Part 2 portion of the study. Patients were analyzed overall, due to a small sample size. Although different Givinostat dose levels were administered, results data are reported only for the "overall" Givinostat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall
Number analyzed (Participants) | 19
score on a scale | -0.2 (2.69)

8. Secondary Outcome: Change From Baseline in Muscular Function After After 24 (Extension 1), 36 (Extension 2), and 52 Months (Extension 3) of Treatment With Givinostat at the Selected Daily Dose Based on the 6-Minute Walk Test
Description: as for outcome 5
Time Frame: At 24, 36, and 52 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Overall: Givinostat was administered as 2 oral doses daily while the child is in fed state.
  Givinostat, oral suspension 10 mg/mL or oral capsules 50 mg, was administered at the dose of 25 mg BID, 37.5 mg BID, and 50 mg BID during Part 1, and 25 mg BID and 37.5 mg BID during Part 2.
  Givinostat oral suspension 10 mg/mL was administered orally at the dose of 25 mg BID or 37.5 mg BID during Extension 1; the dose was modified as per patient's weight during Extensions 2 and 3.
Arm/Group | Overall
Number analyzed (Participants) | 19
meters
  Extension 1 | -80.0 (110.69)
  Extension 2 | -127.0 (110.40)
  Extension 3: number analyzed (Participants) | 18
  Extension 3 | -287.8 (159.47)

9. Secondary Outcome: Change From Baseline in Muscular Function After 24 (Extension 1), 36 (Extension 2), and 52 Months (Extension 3) of Treatment With Givinostat at the Selected Daily Dose Based on the North Star Ambulatory Assessment (NSAA)
Description: as for outcome 6
Time Frame: At 24, 36, and 52 months
Population: The ITT population included all children who were enrolled in the Part 1 portion or entered the Part 2 portion of the study. Patients were analyzed overall due to a small sample size. Although different Givinostat dose levels were administered, results data are reported only for the "overall" Givinostat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall
Number analyzed (Participants) | 18
score on a scale
  Extension 1 | -5.2 (5.06)
  Extension 2 | -7.4 (5.90)
  Extension 3 | -15.2 (7.83)

10. Secondary Outcome: Change From Baseline in Muscular Function After 24 (Extension 1), 36 (Extension 2), and 52 Months (Extension 3) of Treatment With Givinostat at the Selected Daily Dose Based on the Performance of Upper Limb (PUL)
Description: The PUL (version 1.2) was used to assess the change in motor performance of the upper limb over time in patients with Becker and Duchenne muscular dystrophy, from when they are still ambulant, until they loose all arm function when non-ambulant.
  The revised version of the PUL included 22 items taking. These include one entry item to define the starting functional level, and 21 items subdivided into:
  * shoulder level (Question B to E; minimum score 0 and maximum score 16)
  * elbow level (Question F to N; minimum score 0 and maximum score 34)
  * distal level dimension (Question O to V; minimum score 0 and maximum score 24) The total score is calculated by the sum of all the scores of the three subscales (total score range: 0-74) (scores from Question A "entry item" did not contribute). For all items, the higher the score, the better the outcome.
Time Frame: At 24, 36, and 52 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall
Number analyzed (Participants) | 19
score on a scale
  Extension 1: number analyzed (Participants) | 18
  Extension 1 | -0.2 (2.71)
  Extension 2: number analyzed (Participants) | 18
  Extension 2 | -0.2 (2.75)
  Extension 3: number analyzed (Participants) | 18
  Extension 3 | -4.4 (6.09)

11. Secondary Outcome: Number of Children Experiencing Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Type and Severity of TEAEs
Description: Summary of Treatment-emergent Adverse Events (TEAE) Reporting from Baseline to the End of Extension 3 (Month 52). In the analysis were included: Any TEAE, Any treatment-related TEAE, Any mild or moderate or severe TEAE, Any life-threatening or disabling TEAE, Any TEAE resulting in death, any serious adverse event, and Any TEAE resulting in study discontinuation.
Time Frame: Part 1, Part 2, and Extensions 1, 2, and 3
Population: The safety population included all children who received any investigational product. Although different Givinostat dose levels were administered, results data are reported only for the "overall" Givinostat population. During the extension period the dosage was adjusted by patient weight
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 20
participants
  TEAEs | 20
  Any treatment-related TEAE | 20
  Any mild TEAE | 20
  Any moderate TEAE | 16
  Any severe TEAE | 9
  Any life-threatening or disabling TEAE | 1
  Ant TEAE resulting in death | 0
  Any SAE | 8
  Any TEAE resulting in study discontinuation | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were assessed throughout the study: in Part 1 (screen, weeks 0, 1, 2, 3, 4, 5); Part 2 (months 0, 1, 2, 3, 4.5, 6, 7.5, 9, 10.5,12); Extension 1 (months 14,16,18, 20, 22, 24, FU); Extension 2 (months 26,28, 30,32, 34, 36, FU); Extension 3 (months 40, 44, 48, 52, FU). Extensions 1, 2 and 3 together represent Part 3 of the study.
Description: TEAEs by Primary System Organ Class, Preferred Term, and Relationship to Study Drug are reported for each dose separately in Part 1 and Part 2 of the study (i.e. Part 1 25.0 mg, Part 1 37.5 mg, Part 1 50 mg; Part 2 25.0 mg, Part 2 37.5 mg) and are reported to represent all participants and all parts of this study including the extension period altogether (i.e. Part 1 + Part 2 + Extensions 1, 2, and 3). Adverse events were not assessed by dose nor separately for the extension period.
Groups:
- Part 1 - 25 mg; Part 1 - 50 mg; Part 1 - 37.5 mg: The safety population included all children who received any investigational product. The dose level under which the patient was analyzed was the dose of investigational product that was actually received.
  19 patients were included in the safety population of Part 1.
- Part 2 - 37.5 mg; Part 2 - 25 mg: The safety population included all children who received any investigational product. The dose level under which the patient was analyzed was the dose of investigational product that was actually received.
  19 patients were included in the safety population of Part 2.
- Overall (Part 1 + Part 2 + Extensions 1, 2, 3 ): The safety population included all children who received any investigational product. The dose level under which the patient was analyzed was the dose of investigational product that was actually received.
  19 patients were included in the safety population of Part 1 and 19 patients were included in the safety population of Part 2.
  In all Extensions, the Safety Analysis Population was set up to 20 patients (100%), including all patients who received any investigational product.
Arm/Group | Part 1 - 25 mg | Part 1 - 50 mg | Part 1 - 37.5 mg | Part 2 - 37.5 mg | Part 2 - 25 mg | Overall (Part 1 + Part 2 + Extensions 1, 2, 3 )
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/12 | 0/7 | 0/19 | 0/12 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/12 | 0/7 | 1/19 | 1/12 | 8/20
Other Adverse Events (participants affected / at risk) | 3/4 | 12/12 | 6/7 | 19/19 | 12/12 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - 25 mg (N=4) | Part 1 - 50 mg (N=12) | Part 1 - 37.5 mg (N=7) | Part 2 - 37.5 mg (N=19) | Part 2 - 25 mg (N=12) | Overall (Part 1 + Part 2 + Extensions 1, 2, 3 ) (N=20)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataracts (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femural fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lower limb fracture (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - 25 mg (N=4) | Part 1 - 50 mg (N=12) | Part 1 - 37.5 mg (N=7) | Part 2 - 37.5 mg (N=19) | Part 2 - 25 mg (N=12) | Overall (Part 1 + Part 2 + Extensions 1, 2, 3 ) (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Left ventricular dilatation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular disfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Delayed puberty (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Secondary adrenocartical insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Lens discoloration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lenticular opacity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 2 (3) | 5 (6) | 0 (0) | 11 (19)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (8) | 3 (4) | 9 (23) | 6 (14) | 15 (66)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 8 (11)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 9 (20)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 9 (14)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 8 (9)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Legament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Legament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 5 (7)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord injury sacral (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 3 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 13 (18) | 5 (7) | 13 (39)
White blood cell count decreased (Investigations) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 4 (7)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 7 (8)
Hypertryglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (5)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 4 (6)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-08-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT01761292/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT01761292/SAP_001.pdf